CLINICAL TRIAL: NCT02983461
Title: Use of Sildenafil for Treatment of Urinary Incontinence
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-0121
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; pelvic floor dysfunction
MeSH Terms: conditions — Urinary Incontinence | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Double Blind Placebo 3 times a day for 10 weeks.
  Interventions: Drug: Placebo
- Sildenafil (Active Comparator): Double Blind Sildenafil, 20mg x 3 times a day, 10 weeks.
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — Sildenafil, 20mg x 3 times a day for 10 weeks
  Arms: Sildenafil
Drug: Placebo — Placebo oral tablet, 3 times a day for 10 weeks
  Arms: Placebo

SUMMARY:
The investigators goal is to develop medical treatments for stress/mixed urinary incontinence. Sildenafil has been shown to improve blood flow as well as muscle mass and strength and to decrease muscle fatigue. The investigators believe that it will improve muscular atrophy in the pelvic floor, thus improving symptoms of urinary incontinence related to pelvic floor dysfunction.

DETAILED DESCRIPTION:
Aim: To determine the effect of sildenafil on urinary incontinence.

1. Episodes of urinary incontinence will be recorded using a 3 day bladder diary.
2. Quantitative assessment of urinary incontinence will be performed at baseline and after treatment using a Pad Test.
3. Muscle strength will be assessed through use of a perineometer.
4. To evaluate macrocirculatory blood flow in pelvic organs, women will be assessed with noninvasive imaging before and after randomization to sildenafil.
5. Secondary outcomes will include evaluation of muscle and vaginal mucosal thickness.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal females, 50-80 years of age, at the time of consent
* Have stress or mixed urinary incontinence, with at least 3 episodes/week
* Willing and able to comply with study procedures
* Willing and able to provide written informed consent

Exclusion Criteria:

* Significant heart, liver, kidney, pulmonary, blood, autoimmune or peripheral vascular disease (history of Hashimoto's thyroiditis is not exclusionary if stable and thyroid replacement is being administered. Thyroid testing will be performed at screening and as needed during study visits. )
* Systolic blood pressure <100 or >150, diastolic blood pressure <60 or >90 after repeated evaluation with proper cuff. This range is smaller than the acceptable range stated in the prescribing information for sildenafil (>90/50 and <170/110)
* Diabetes mellitus or other untreated endocrine disease
* Active cancer
* Currently using and planning to continue use of urinary incontinence medications during study period
* BMI > 40
* HIV, Hepatitis B, or Hepatitis C
* Use of systemic nitrates, anabolic steroids or corticosteroids in the past 6 months
* Use of alpha blockers
* Any medical condition that, in the opinion of the investigator, would place the subject at increased risk for participation.
* Known allergic reaction to any agent under investigation or required by the protocol.
* History of prior non-compliance or the presence or history of psychiatric condition (including drug or alcohol addiction) that would, in the opinion of the investigator, make it difficult for the subject to comply with the study procedures or follow the investigators instructions.
* Females who are pregnant or lactating.

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-03-10 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Urinary Incontinence as measured by Pad Test | 10 weeks
  Pad tests quantitatively measures urine leakage

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen L Vincent, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States